CLINICAL TRIAL: NCT02631096
Title: A Phase 2a Single-Blind, Randomized, Placebo-Controlled Study Evaluating the Safety, Anti Viral Activity, and Pharmacokinetics of ARB-001467 in Non Cirrhotic, HBeAg Negative and Positive Subjects With Chronic HBV Infection Receiving Nucleos(t)Ide Analogue Therapy
Brief Title: Study of ARB-001467 in Subjects With Chronic HBV Infection Receiving Nucleos(t)Ide Analogue Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARB-001467-002
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single Blind (Subject) in cohort 1-3, Open label in Cohort 4
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 0.2 mg/kg ARB-001467 or Placebo (Experimental): HBeAg-negative subjects randomized 3:1 to receive ARB-001467 at 0.2 mg/kg versus placebo once a month for 3 months
  Interventions: Drug: ARB-001467; Other: Placebo
- 0.4 mg/kg ARB-001467 or Placebo (Experimental): HBeAg-negative subjects randomized 3:1 to receive ARB-001467 at 0.4 mg/kg versus placebo once a month for 3 months
  Interventions: Drug: ARB-001467; Other: Placebo
- ARB-001467 or Placebo (Experimental): HBeAg-positive subjects randomized 3:1 to receive ARB-001467 at 0.4 mg/kg versus placebo once a month for 3 months
  Interventions: Drug: ARB-001467; Other: Placebo
- 0.4 mg/kg ARB-001467 (Experimental): HBeAg-negative subjects receive ARB-001467 at. 0.4 mg/kg (open label) bi-weekly for 5 treatments and then subjects with HBsAg ≤1000 IU/mL AND ≥1.0 log10 decrease from baseline at Day 71 will continue monthly dosing through 48 weeks
  Interventions: Drug: ARB-001467

INTERVENTIONS:
Drug: ARB-001467 — An IV infusion of ARB-001467
Other: Placebo — An IV infusion of placebo
  Other Names: 0.9% sodium chloride
  Arms: 0.2 mg/kg ARB-001467 or Placebo; 0.4 mg/kg ARB-001467 or Placebo; ARB-001467 or Placebo

SUMMARY:
The study is a phase 2a, single blind, randomized, placebo controlled, study evaluating the safety, anti-viral activity, and pharmacokinetics (PK) following multiple doses of intravenous ARB-001467

DETAILED DESCRIPTION:
Approximately 24 subjects will be enrolled in three cohorts: two cohorts of HBeAg-negative subjects and one cohort of HBeAg-positive subjects and 12 HbeAg-negative subjects will be enrolled in cohort 4. All subjects will be non-cirrhotic, with chronic hepatitis B virus (HBV) infection, and will have been receiving nucleos(t)ide-analogue (NA) therapy with entecavir or tenofovir for at least 12 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Documented chronic HBV infection for ≥12 months prior to Screening Visit.
* Quantitative HBsAg ≥1000 IU/mL at the Screening Visit.
* Subjects currently receiving entecavir and/or tenofovir for ≥12 months and HBV DNA undetectable.

Key Exclusion Criteria:

* Known co-infection with HIV, hepatitis C virus, and hepatitis D virus.
* Receiving or planning to receive systemic immunosuppressive medications during the study or ≤2 months prior to the first dose of study treatment.
* Receiving or planning to receive interferon during the study or ≤12 months prior to the first dose of study treatment.
* Significant immunosuppression from, but not limited to immunodeficiency conditions such as common variable hypogammaglobulinemia.
* Clinical diagnosis of substance abuse with alcohol, narcotics, or cocaine ≤12 months prior to the Screening Visit.
* Any known pre-existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2018-05-18 (Actual); Study Completion 2018-05-18 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent SAEs, discontinuations due to AEs, and laboratory abnormalities, by cohort, through 28 days after the last infusion of study treatment. | 28 days post last infusion
  To evaluate the safety and tolerability of multiple doses of ARB-001467 in HBeAg-negative and HBeAg-positive subjects with chronic Hepatitis B virus infection who are receiving nucleos(t)ide analogue therapy

SECONDARY OUTCOMES:
Evaluate ARB-001467 Maximum plasma concentration (Cmax) at multiple time points from baseline through Day 85; 28 days after the last infusion of study treatment (cohort 1-3) and Week 36 (Cohort 4). | Up to 36 Weeks
  To evaluate the pharmacokinetics of multiple doses of ARB-001467 in subjects with chronic HBV infection.
Evaluate ARB-001467 Time to maximum plasma concentration (Tmax) at multiple time points from baseline through Day 85; 28 days after the last infusion of study treatment (cohort 1-3) and Week 36 (Cohort 4). | Up to 36 Weeks
  To evaluate the pharmacokinetics of multiple doses of ARB-001467 in subjects with chronic HBV infection.
Evaluate ARB-001467 Area under the plasma concentration-time curve from the start of infusion to the last measurable concentration (AUC0-t) at multiple time points from baseline through Day 85 (cohort 1-3) and Week 36 (Cohort 4). | Up to 36 Weeks
  To evaluate the pharmacokinetics of multiple doses of ARB-001467 in subjects with chronic HBV infection.
Evaluate additional parameters for ARB-001467 from plasma concentration-time curve from start of infusion and extrapolated to infinity (AUC0-t), inf) partial, AUCs, T1/2, volume of distribution (VD) and clearance (CL) -baseline through Day 85 or Week 36. | Up to 36 Weeks
  To evaluate the pharmacokinetics of multiple doses of ARB-001467 in subjects with chronic HBV infection.
Evaluate antiviral activity of ARB 001467 for up to 72 weeks after the first dose of study treatment. | Up to 18 months
  The proportion of subjects in each dose level cohort with ≥0.5 log10 HBsAg decrease from baseline at EOS, and for these subjects, the changes from baseline (expressed as percentage and log10 change) in the following virologic markers will be assessed throughout the study:
  * Quantitative HBV surface antigen (HBsAg)
  * Quantitative HBV surface antibody (HBsAb)
  * Quantitative HBV DNA and HBV-RNA (viral load)
  For the HBeAg positive cohort only:
  - Quantitative HBV e antigen (HBeAg)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Mendez, MD, PhD, Study Chair — Arbutus Biopharma Corporation
Locations (4):
- Australia (3):
  - Monash Health, Gastroenterology and Hepatology, Clayton, Victoria
  - The Alfred, Gastroenterology and Hepatology, Melbourne, Victoria
  - Linear Clinical Research Ltd, Nedlands, Western Australia
- Auckland Clinical Studies Ltd, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Undecided